CLINICAL TRIAL: NCT05846685
Title: Preventing Future Falls in Older Adult ED Patients: Evaluating the Implementation and Effectiveness of a Novel Automated Screening and Referral Intervention - Patient Perspectives
Brief Title: Patient Perspectives of an Automated Falls-Risk Screening and Referral Tool in the Emergency Department (ED)
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2021-0744; 1K08HS024558 (AHRQ); 1R18HS027735 (AHRQ); SMPH/EMERG MED (Other: UW Madison)
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Falls-Risk
Keywords: Machine Learning; Computer Decision Support; Human Factors Engineering; Qualitative Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ED Patients Scheduled and Completed Falls Clinic Visit: Patients age 65 and Older identified by the automated system as being high-risk of future falls, and subsequently referred to the UW Health Mobility and Falls Clinic by the ED provider at discharge
  Interventions: Other: Patient Phone Interviews
- ED Patients Declined or Did Not Complete Falls Clinic Visit: Patients age 65 and Older identified by the automated system as being high-risk of future falls, and subsequently referred to the UW Health Mobility and Falls Clinic by the ED provider at discharge
  Interventions: Other: Patient Phone Interviews
- ED Patients Likely to be Discharged: Patients aged 65 and older who are in the emergency department and likely to be discharged.
  Interventions: Other: Patient In Person Interviews

INTERVENTIONS:
Other: Patient Phone Interviews — Collecting perceptions about automated falls-risk screening and referral tool
  Groups: ED Patients Declined or Did Not Complete Falls Clinic Visit; ED Patients Scheduled and Completed Falls Clinic Visit
Other: Patient In Person Interviews — Interviews will be aimed at collecting patient input necessary to adapt the design of the intervention at these sites.
  Groups: ED Patients Likely to be Discharged

SUMMARY:
The purpose of the overall study to evaluate implementation-related outcomes of a falls-risk clinical decision support (CDS) system using patient electronic health records (EHR) data to automatically screen and identify older adult ED patients at high risk of future falls and allowing ED clinicians to place referral orders to the UW Health Mobility and Falls clinic. This CDS tool has already been implemented at the UWHC ED, and will be additionally implemented at The American Center and Swedish American Hospital EDs (all QI initiatives) over the next two years. This study involves engaging a sample of referred patients from each site to gather their perspectives on the delivery of the referral in the ED, their experiences in making and completing appointments at the Falls Clinic (if applicable), and perceived benefits of the intervention overall.

DETAILED DESCRIPTION:
The aim of this study is to assess perceptions and implementation-related outcomes for the automated screening and referral tool based upon the experiences of older adult patients receiving the referral (or who could be eligible for the referral) at each of the three ED sites, including identifying reasons why some referred patients do not schedule or attend appointments as a result of the referral order.

Phone interviews will be conducted with a minimum of 12 referred patients per each of the 3 ED sites, approximately half of whom scheduled and completed a Falls Clinic visit, and half whom declined or did not complete an appointment. Interview questions include a mix of verbally-delivered Likert-type rating scales and open-ended questions evaluating their experience of the referral process (e.g., verbal communication, written information received), appropriateness of the CDS screening tool, and perceived value of the intervention for preventing falls.

Additionally, in person interviews will be conducted with a minimum of 10 patients each at the American Center and Swedish American Hospital sites prior to implementation of the intervention at these sites. These will be conducted among patients aged 65 and older who are in the emergency department and likely to be discharged. These interviews will be aimed at collecting patient input necessary to adapt the design of the intervention at these sites. Interview questions will include open-ended questions evaluating the perceived value of the the intervention for preventing falls as well as potential barriers and facilitators to completing the intervention at these sites. Interviews will be conducted by ED staff trained and experienced in research data collection in the ED to minimize interruption of clinical workflows. In consultation with provider teams, interviewers will time interviews to avoid clinical interventions, and will pause research activities while any clinical care is taking place.

ELIGIBILITY:
Inclusion Criteria:

* ED patients identified by the automated system as being high-risk of future falls, and subsequently referred to the UW Health Mobility and Falls Clinic by the ED provider at discharge.
* English-speaking
* Reliable access to a working telephone and can accept incoming phone calls
* For In-person interviews in the ED:

  * ED patients age 65 and older in the emergency department for any reason who are identified as likely to be discharged by their clinical team.

Exclusion Criteria:

* Incarcerated or in police custody
* Lacks capacity to consent
* Unable to hear or speak on the telephone, even with the use of assistive devices

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: ED patients age 65 or older
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Qualitative Measure to Summarize Reasons Patients Did Not Schedule or Attend Appointments Based on Referral | up to 30 months
  Participant responses will be coded to identify themes. Participant counts will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Brian W Patterson, MD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Swedish American Emergency Department, Rockford, Illinois
  - The American Center Emergency Department, Madison, Wisconsin
  - UWHC Emergency Department, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No